CLINICAL TRIAL: NCT01266850
Title: Safety and Immunogenicity of Sequential Rotavirus Vaccine Schedules With RotaTeq® and Rotarix®
Brief Title: Safety and Immunogenicity of Sequential Rotavirus Vaccine Schedules
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-0017; N01AI80006C
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Results first posted 2014-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-09

CONDITIONS: Rotavirus Infection
Keywords: vaccine, rotavirus, gastroenteritis, infants
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis | interventions — RIX4414 vaccine; RotaTeq

ARMS (5):
- Group 1, RotaTeq® x 3 (Active Comparator): 2, 4 and 6 months of age: RotaTeq®
  Interventions: Biological: RotaTeq®
- Group 5, Rotarix®, RotaTeq® x2 (Experimental): 2 months of age: Rotarix®; 4 and 6 months of age: RotaTeq®
  Interventions: Biological: Rotarix®; Biological: RotaTeq®
- Group 4, Rotarix® x 2 (Active Comparator): 2 and 4 months of age: Rotarix®
  Interventions: Biological: Rotarix®
- Group 2, RotaTeq®, Rotarix® x 2 (Experimental): 2 months of age: RotaTeq®; 4 and 6 months of age: Rotarix®
  Interventions: Biological: Rotarix®; Biological: RotaTeq®
- Group 3, RotaTeq® x 2, Rotarix® (Experimental): 2 and 4 months of age: RotaTeq®; 6 months of age: Rotarix®
  Interventions: Biological: Rotarix®; Biological: RotaTeq®

INTERVENTIONS:
Biological: Rotarix® — Each 1-mL dose of Rotarix® contains a suspension of at least 10^6 median Cell Culture Infective Dose (CCID50) of live, attenuated human G1P rotavirus after reconstitution. The lyophilized vaccine contains amino acids, dextran, Dulbecco's Modified Eagle Medium (DMEM), sorbitol, and sucrose. The liquid diluent contains calcium carbonate, sterile water, and xanthan. The diluent includes an antacid component (calcium carbonate) to protect the vaccine during passage through the acid environment of the stomach. Rotarix® contains no preservatives. Once reconstituted, the vaccine will appear white and turbid.
  Arms: Group 2, RotaTeq®, Rotarix® x 2; Group 3, RotaTeq® x 2, Rotarix®; Group 4, Rotarix® x 2; Group 5, Rotarix®, RotaTeq® x2
Biological: RotaTeq® — 2-mL ready-to-use oral solution of live reassortant rotaviruses, containing G1, G2, G3, G4, and P1A, which contains a minimum of 2.0 to 2.8 x 10^6 infectious units (IU) per individual reassortant dose, depending on the serotype, and not greater than 116 x 10^6 IU per aggregate dose. The buffered stabilizer solution contains sucrose, sodium citrate, sodium phosphate monobasic monohydrate, sodium hydroxide, polysorbate 80, cell culture media, and trace amounts of fetal bovine serum. RotaTeq® contains no preservatives. RotaTeq® is a pale yellow clear liquid that may have a pink tint.
  Arms: Group 1, RotaTeq® x 3; Group 2, RotaTeq®, Rotarix® x 2; Group 3, RotaTeq® x 2, Rotarix®; Group 5, Rotarix®, RotaTeq® x2

SUMMARY:
Rotavirus, sometimes called the "stomach flu," is the most common cause of severe diarrhea in children. Vaccines can prevent many types of infections and work by causing the body to make proteins called antibodies that fight infection. For some vaccines, more than one vaccination is needed so that the body will make enough antibodies to fight infection. The vaccines (RotaTeq® or Rotarix® oral vaccines) given in this study are recommended for infants by the Centers for Disease Control and Prevention (CDC) Advisory Committee on Immunization Practices (ACIP). These vaccines require either 2 or 3 vaccinations to be effective. Healthy infants between 6 weeks and 14 weeks, 6 days of age at Visit 1 will participate for about 10-12 months. Study procedures include reaction assessment and blood sample.

DETAILED DESCRIPTION:
Rotavirus is the most common cause of severe gastroenteritis among children. The purpose of the proposed study is to determine the non-inferiority and safety of the 2 licensed rotavirus vaccines when both are administered to the same child during sequential vaccinations. Both Rotarix® and RotaTeq® vaccines have been evaluated for safety and efficacy in placebo-controlled trials with more than 70,000 infants each and it is likely that both vaccines delivered in various combinations will be safe and effective. Since RotaTeq® was licensed in the United States (US) in 2006, approximately 6 million doses have been administered in the US. In addition, Rotarix® has been licensed in over 100 nations worldwide and has been delivered to many children in Latin America where it has been recommended for universal vaccination for over 2 years. Now both RotaTeq® and Rotarix® are licensed in the US, and it is expected that health care providers will administer both vaccines. A 3-dose regimen is recommended for RotaTeq® and a 2-dose regimen for Rotarix®. From previous experience, it is likely that one of the vaccines may become unavailable for some period or pediatric offices may switch from one vaccine to the other. Thus, it is probable that mixed schedules will be administered to infants. The primary objective is to determine if the proportion of seroresponders in the sequential mixed rotavirus vaccine groups (RotaTeq® and Rotarix®) is non-inferior to the proportion of seroresponders in the recommended schedule of the single vaccine alone group. Secondary Objectives are: to determine the neutralizing rotavirus antibody responses to the most common rotavirus serotypes (G1-G4 and G9) at 3-6 weeks after the last vaccination for both the sequential, mixed rotavirus vaccine schedule and the single rotavirus vaccine recommended schedule; and to determine if sequential mixed rotavirus vaccine schedules are safe with no statistically significant increase in fever, diarrhea, vomiting, or intussusception in the mixed schedule groups when compared with the recommended schedule of the single vaccine alone group. Normal healthy full-term infants who are scheduled to receive their routine infant immunizations and who are at least 6 weeks of age and no more than 14 weeks, 6 days of age at Visit 1 will be recruited from their primary care clinic. Infants will be randomized (open label) to one of 5 different rotavirus vaccine study groups. Two study groups will be administered the standard RotaTeq® or Rotarix® vaccines as 3 and 2 doses, respectively, and 3 study groups will be administered mixed sequences of RotaTeq® and Rotarix® given as 3 doses. All rotavirus vaccines will be administered concurrently with the other routinely administered childhood vaccines. Parents/legal guardians will be given a memory aid and a thermometer, and asked to record any suspected fever (with measured temperature documented) or adverse events for Days 1-8 after vaccination. At approximately 1 week after vaccination, study personnel will contact the parents/legal guardians, review the completed memory aid, and record the findings on the case report form. Blood for immunogenicity testing will be obtained 3-6 weeks after the last dose of vaccine. For the four 3-dose rotavirus vaccine study groups, blood will be obtained at approximately 7 months of age (3-6 weeks after the last rotavirus vaccine dose). For the single Rotarix® vaccine study group, blood will be obtained at approximately 5 months of age (3-6 weeks after the last dose of Rotarix® vaccine). The primary analysis will be based on rates of induction of anti-rotavirus serum immunoglobulin (Ig) A in the 5 study groups 3-6 weeks

ELIGIBILITY:
Inclusion Criteria:

* Male or female infants who are at least 6 weeks of age and no more than 14 weeks, 6 days of age at Visit 1.
* Parent(s)/legal guardian(s) have signed informed consent documents.
* Children who will be available for the entire study period and whose parents/legal guardians can be reached by telephone.
* Healthy infants as determined by medical history and by a baseline physical examination with no clinically significant abnormal findings within 14 days before the first dose.
* Parents/legal guardians able to complete all relevant study procedures during study participation.

Exclusion Criteria:

* Any clinically significant history of gastrointestinal disease including abdominal surgery or liver disease or other serious medical conditions as determined by the site investigator.
* Any history of immunodeficiency in the infant (e.g., the infant is known to be human immunodeficiency virus (HIV) positive, to have hypogammaglobulinemia, or to have an underlying malignancy), or any infant with any unvaccinated household contact who is immunocompromised such as:

  * Any malignancies or are otherwise immunocompromised;
  * Primary immunodeficiency; or
  * Receiving immunosuppressive therapy.
* Known sensitivity to any vaccine components, such as latex in the Rotarix® applicator.
* Previous receipt of a rotavirus vaccine.
* Acute illness at the time of vaccine administration, such as any of the following within the past 48 hours:

  1. Axillary temperature of 100.4 degrees Fahrenheit or higher, or
  2. More than 3 grossly watery stools, or
  3. Any episodes of vomiting (forceful expulsion of partially digested milk/food). Infants with previous diagnoses of gastroesophageal reflux whose regurgitation episodes have not changed in the 48-hour period prior to the first vaccination may be enrolled.

If these symptoms clear within 48 hours and the subject meets the other inclusion/exclusion criteria, then the subject may be enrolled.

* The subject is currently participating in a study that involves an experimental agent (vaccine, drug, biologic, device, blood product, or medication) or has received an experimental agent within 1 month prior to enrollment in this study, or expects to receive another experimental agent during participation in this study.
* Less than 37 weeks gestation at birth.
* Receipt of blood and/or blood products (including immunoglobulin) within 4 weeks before vaccine administration.
* Receipt of live vaccine within the past 30 days or a nonreplicating, inactivated, or subunit vaccine within the last 14 days, although planned licensed trivalent inactivated influenza vaccine that may be administered to children over 6 months of age during a routine clinic visit is permitted and would not be exclusionary.
* The subject has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 6 Weeks to 14 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1384 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Kaiser Permanente Vaccine Study Center, Oakland, California
  - Children's Hospital & Research Center Oakland - Primary Care Clinic, Oakland, California
  - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - University of Iowa - Vaccine Research & Education Unit, Iowa City, Iowa
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Children's Mercy Hospital and Clinics - Infectious Diseases, Kansas City, Missouri
  - Duke Translational Medicine Institute - Clinical Vaccine Unit, Durham, North Carolina
  - Primary Physicians Research Inc. - Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee
  - The University of Texas Medical Branch - Sealy Center for Vaccine Development (SCVD), Galveston, Texas
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Group Health Research Institute - Seattle, Seattle, Washington
  - Seattle Children's Hospital - Infectious Diseases, Seattle, Washington

REFERENCES:
- [Derived] Libster R, McNeal M, Walter EB, Shane AL, Winokur P, Cress G, Berry AA, Kotloff KL, Sarpong K, Turley CB, Harrison CJ, Pahud BA, Marbin J, Dunn J, El-Khorazaty J, Barrett J, Edwards KM; VTEU Rotavirus Vaccine Study Work Group. Safety and Immunogenicity of Sequential Rotavirus Vaccine Schedules. Pediatrics. 2016 Feb;137(2):e20152603. doi: 10.1542/peds.2015-2603. Epub 2016 Jan 28. PMID 26823540

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy males and females age 6-14 weeks, recruited from the communities at large around the clinical sites. Participants were enrolled and vaccinated between 24MAR2011 and 08APR2013.
Groups:
- Group 1: RotaTeq, RotaTeq, RotaTeq: Participants received RotaTeq® orally at 2, 4 and 6 months of age.
- Group 2: RotaTeq, Rotarix, Rotarix: Participants received RotaTeq® orally at 2 months of age, followed by Rotarix® orally at 4 and 6 months of age.
- Group 3: RotaTeq, RotaTeq, Rotarix: Participants received RotaTeq® orally at 2 and 4 months of age, followed by Rotarix® orally at 6 months of age.
- Group 4: Rotarix, Rotarix: Participants received Rotarix® orally at 2 and 4 months of age.
- Group 5: Rotarix, RotaTeq, RotaTeq: Participants received Rotarix® orally at 2 months of age, followed by RotaTeq® orally at 4 and 6 months of age.
Period: Overall Study
Arm/Group | Group 1: RotaTeq, RotaTeq, RotaTeq | Group 2: RotaTeq, Rotarix, Rotarix | Group 3: RotaTeq, RotaTeq, Rotarix | Group 4: Rotarix, Rotarix | Group 5: Rotarix, RotaTeq, RotaTeq
Started | 242 | 248 | 238 | 329 | 327
Received Second Vaccine | 231 | 233 | 227 | 311 | 307
Received Third Vaccine | 221 | 221 | 217 | 0 | 299
Completed | 212 | 212 | 214 | 301 | 297
Not Completed | 30 | 36 | 24 | 28 | 30
Not completed — Lost to Follow-up | 19 | 19 | 13 | 13 | 12
Not completed — Withdrawal by Subject | 8 | 9 | 6 | 9 | 12
Not completed — Physician Decision | 3 | 6 | 4 | 4 | 3
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Site Closure | 0 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Population for baseline analysis includes all participants who were enrolled, randomized, and received at least the first vaccination.
Groups:
- Group 1: RotaTeq, RotaTeq, RotaTeq: Participants received 2-mL RotaTeq® orally at 2, 4 and 6 months of age.
- Group 2: RotaTeq, Rotarix, Rotarix: Participants received 2-mL RotaTeq® orally at 2 months of age, followed by 1-mL Rotarix® orally at 4 and 6 months of age.
- Group 3: RotaTeq, RotaTeq, Rotarix: Participants received 2-mL RotaTeq® orally at 2 and 4 months of age, followed by 1-mL Rotarix® orally at 6 months of age.
- Group 4: Rotarix, Rotarix: Participants received 2-mL Rotarix® orally at 2 and 4 months of age.
- Group 5: Rotarix, RotaTeq, RotaTeq: Participants received 2-mL Rotarix® orally at 2 months of age, followed by 1-mL RotaTeq® orally at 4 and 6 months of age.
- Total: Total of all reporting groups
Arm/Group | Group 1: RotaTeq, RotaTeq, RotaTeq | Group 2: RotaTeq, Rotarix, Rotarix | Group 3: RotaTeq, RotaTeq, Rotarix | Group 4: Rotarix, Rotarix | Group 5: Rotarix, RotaTeq, RotaTeq | Total
Number analyzed (Participants) | 242 | 248 | 238 | 329 | 327 | 1384
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 9.2 (1.4) | 9.1 (1.2) | 9.2 (1.2) | 9.1 (1.2) | 9.2 (1.4) | 9.2 (1.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 242 | 248 | 238 | 329 | 327 | 1384
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 112 | 125 | 176 | 149 | 686
  Male | 118 | 136 | 113 | 153 | 178 | 698
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 1 | 3
  Asian | 5 | 4 | 4 | 12 | 8 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 4 | 1 | 1 | 0 | 6
  Black or African American | 60 | 57 | 52 | 80 | 81 | 330
  White | 143 | 143 | 139 | 199 | 195 | 819
  More than one race | 30 | 35 | 37 | 33 | 41 | 176
  Unknown or Not Reported | 3 | 5 | 4 | 4 | 1 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 49 | 45 | 52 | 67 | 254
  Not Hispanic or Latino | 201 | 199 | 193 | 277 | 260 | 1130
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 242 | 248 | 238 | 329 | 327 | 1384

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Developing a Serum Anti-rotavirus Immunoglobulin (Ig) A Titer of 20 or Greater in the WC3 IgA Assay
Description: Blood was collected from all participants at the follow up visit 3-6 weeks after the last vaccination for testing in the ELISA assay to determine the anti-rotavirus IgA antibody titer. A participant met the threshold of a positive response if the post vaccination anti-rotavirus IgA antibody titer was 20 or greater.
Time Frame: 3-6 weeks after the last vaccination
Population: The per protocol analysis population includes participants who met all inclusion and exclusion criteria, received all scheduled study vaccinations, and who contributed post-vaccination blood samples for testing for which valid results were reported.
Measure: Number; unit: participants
Arm/Group | Group 1: RotaTeq, RotaTeq, RotaTeq | Group 2: RotaTeq, Rotarix, Rotarix | Group 3: RotaTeq, RotaTeq, Rotarix | Group 4: Rotarix, Rotarix | Group 5: Rotarix, RotaTeq, RotaTeq
Number analyzed (Participants) | 206 | 206 | 194 | 287 | 280
participants | 186 | 182 | 175 | 191 | 261

2. Primary Outcome: Number of Participants Developing a Serum Anti-rotavirus Immunoglobulin (Ig) A Titer of 20 or Greater in the 89-12 IgA Assay
Description: Blood was collected from all participants at the follow up visit 3-6 weeks after the last vaccination for testing in the ELISA 89-12 assay to determine the anti-rotavirus IgA antibody titer. A participant met the threshold of a positive response if the post vaccination anti-rotavirus IgA antibody titier was 20 or greater.
Time Frame: 3-6 weeks after the last vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1: RotaTeq, RotaTeq, RotaTeq | Group 2: RotaTeq, Rotarix, Rotarix | Group 3: RotaTeq, RotaTeq, Rotarix | Group 4: Rotarix, Rotarix | Group 5: Rotarix, RotaTeq, RotaTeq
Number analyzed (Participants) | 206 | 207 | 193 | 287 | 280
participants | 159 | 184 | 165 | 219 | 256

3. Secondary Outcome: GMT of Neutralizing Rotavirus Antibody to the Most Common Rotavirus Serotypes (G1-G4 and G9)
Description: Blood was collected from all participants at the follow up visit 3-6 weeks after the last vaccination for testing in the neutralizing antibody assay against the most common rotavirus serotypes, G1-G4 and G9. Antigen-specific geometric mean titers (GMT) for each group were calculated along with the 95% confidence intervals.
Time Frame: 3-6 weeks after the last dose of vaccine.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: RotaTeq, RotaTeq, RotaTeq | Group 2: RotaTeq, Rotarix, Rotarix | Group 3: RotaTeq, RotaTeq, Rotarix | Group 4: Rotarix, Rotarix | Group 5: Rotarix, RotaTeq, RotaTeq
Number analyzed (Participants) | 206 | 207 | 195 | 287 | 280
titers
  G1P[8] Antigen | 84.5 [68.81 to 103.72] | 93.6 [76.88 to 114.02] | 112.0 [89.68 to 139.84] | 45.3 [39.60 to 51.75] | 96.6 [81.73 to 114.24]
  G2P[4] Antigen | 17.1 [14.54 to 20.11] | 14.5 [12.33 to 17.02] | 17.5 [14.68 to 20.94] | 7.1 [6.51 to 7.76] | 19.3 [16.50 to 22.62]
  G3,P[8] Antigen | 12.9 [11.06 to 15.01] | 16.8 [14.40 to 19.61] | 16.6 [13.91 to 19.83] | 14.0 [12.50 to 15.65] | 22.2 [18.89 to 25.98]
  G4P[6] Antigen | 18.6 [16.08 to 21.63] | 17.7 [15.18 to 20.74] | 21.3 [17.92 to 25.21] | 7.0 [6.49 to 7.59] | 19.0 [16.58 to 21.74]
  G4P[8] Antigen | 26.1 [22.17 to 30.67] | 22.1 [18.77 to 26.01] | 24.9 [21.22 to 29.28] | 8.7 [7.96 to 9.58] | 25.6 [22.28 to 29.39]
  G9P[6] Antigen | 13.1 [11.24 to 15.38] | 13.5 [11.58 to 15.75] | 16.1 [13.37 to 19.37] | 6.8 [6.37 to 7.34] | 14.5 [12.57 to 16.69]

4. Secondary Outcome: Number of Participants Experiencing Solicited Systemic Reactions in the 8 Days After Vaccination
Description: The participants' parent/guardian was given a memory aid to record for 8 days the presence of solicited reactions of fever, diarrhea and vomiting. Fever was considered experienced if the participant was assessed with an axillary temperature of 100.4F or greater on any day in the 8-day period after any vaccination. Diarrhea was considered experienced if the participant had 3 or more looser than normal stools in a day. Vomiting was considered experienced if the participant vomited 2 or more times in a day.
Time Frame: Days 1-8 after each vaccination
Population: All participants who were vaccinated and had reactogenicity data reported are included in the analysis population.
Measure: Number; unit: participants
Arm/Group | Group 1: RotaTeq, RotaTeq, RotaTeq | Group 2: RotaTeq, Rotarix, Rotarix | Group 3: RotaTeq, RotaTeq, Rotarix | Group 4: Rotarix, Rotarix | Group 5: Rotarix, RotaTeq, RotaTeq
Number analyzed (Participants) | 241 | 245 | 236 | 326 | 325
participants
  Fever | 37 | 36 | 31 | 29 | 49
  Diarrhea | 22 | 27 | 17 | 28 | 32
  Vomiting | 23 | 22 | 18 | 17 | 33

5. Secondary Outcome: Number of Participants Experiencing Hematochezia at Any Time During the Study
Description: Hematochezia was defined as any stools that are black and tarry; maroon in color; or frank red blood. At each visit, signs of hematochezia were assessed and the participant's parent/guardian was instructed to contact the clinical site at any time if the participant had evidence of hematochezia.
Time Frame: Day 1 through 6 months after the last vaccination
Population: All participants who were vaccinated are included in the analysis population.
Measure: Number; unit: participants
Arm/Group | Group 1: RotaTeq, RotaTeq, RotaTeq | Group 2: RotaTeq, Rotarix, Rotarix | Group 3: RotaTeq, RotaTeq, Rotarix | Group 4: Rotarix, Rotarix | Group 5: Rotarix, RotaTeq, RotaTeq
Number analyzed (Participants) | 241 | 245 | 236 | 326 | 325
participants | 5 | 3 | 5 | 6 | 13

6. Primary Outcome: Geometric Mean Serum Anti-rotavirus IgA Titer
Description: Blood was collected from all participants at the follow up visit 3-6 weeks after the last vaccination for testing in the ELISA assay to determine the anti-rotavirus IgA antibody titers. The geometric mean titers (GMT) for each group were calculated along with the 95% confidence intervals.
Time Frame: 3-6 weeks after the last dose of vaccine
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: RotaTeq, RotaTeq, RotaTeq | Group 2: RotaTeq, Rotarix, Rotarix | Group 3: RotaTeq, RotaTeq, Rotarix | Group 4: Rotarix, Rotarix | Group 5: Rotarix, RotaTeq, RotaTeq
Number analyzed (Participants) | 206 | 207 | 195 | 287 | 280
titers
  WC3 Assay | 294.03 [231.519 to 373.407] | 215.81 [168.355 to 276.652] | 305.89 [238.614 to 392.130] | 38.06 [31.715 to 45.685] | 256.90 [214.441 to 307.765]
  89-12 Assay | 60.89 [49.355 to 75.121] | 115.72 [94.543 to 141.642] | 104.04 [83.026 to 130.383] | 100.21 [80.582 to 124.629] | 212.52 [173.815 to 259.833]

7. Secondary Outcome: Number of Participants Developing Neutralizing Rotavirus Antibody to Rotavirus Serotypes G1, G2, G4P6 and G9
Description: Blood was collected from all participants at the follow up visit 3-6 weeks after the last vaccination for testing in the ELISA assay to determine the antibody titers to rotavirus serotypes G1, G2, G4P6 and G9. A participant met the threshold of a positive response if the post vaccination antigen-specific antibody titer was 10 or greater.
Time Frame: 3-6 weeks after the last dose of vaccine.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1: RotaTeq, RotaTeq, RotaTeq | Group 2: RotaTeq, Rotarix, Rotarix | Group 3: RotaTeq, RotaTeq, Rotarix | Group 4: Rotarix, Rotarix | Group 5: Rotarix, RotaTeq, RotaTeq
Number analyzed (Participants) | 206 | 207 | 194 | 287 | 280
participants
  G1P[8] Antigen | 187 | 192 | 176 | 260 | 260
  G2P[4] Antigen | 127 | 112 | 116 | 61 | 165
  G4P[6] Antigen | 146 | 136 | 145 | 68 | 195
  G9P[6] Antigen | 110 | 109 | 112 | 71 | 154

8. Secondary Outcome: Number of Participants Developing Neutralizing Rotavirus Antibody to Rotavirus Serotype G3
Description: Blood was collected from all participants prior to vaccination and at the follow up visit 3-6 weeks after the last vaccination for testing in the ELISA assay to determine the antibody titers to rotavirus serotype G3. A participant met the threshold of a positive response if the post vaccination antibody titer was 10 or greater.
Time Frame: 3-6 weeks after the last dose of vaccine.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1: RotaTeq, RotaTeq, RotaTeq | Group 2: RotaTeq, Rotarix, Rotarix | Group 3: RotaTeq, RotaTeq, Rotarix | Group 4: Rotarix, Rotarix | Group 5: Rotarix, RotaTeq, RotaTeq
Number analyzed (Participants) | 205 | 207 | 194 | 287 | 280
participants | 108 | 134 | 111 | 179 | 189

9. Secondary Outcome: Number of Participants Developing Neutralizing Rotavirus Antibody to Rotavirus Serotypes G4P8
Description: Blood was collected from all participants at the follow up visit 3-6 weeks after the last vaccination for testing in the ELISA assay to determine the antibody titers to rotavirus serotype G4P8. A participant met the threshold of a positive response if the post vaccination antibody titer was 10 or greater.
Time Frame: 3-6 weeks after the last dose of vaccine.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1: RotaTeq, RotaTeq, RotaTeq | Group 2: RotaTeq, Rotarix, Rotarix | Group 3: RotaTeq, RotaTeq, Rotarix | Group 4: Rotarix, Rotarix | Group 5: Rotarix, RotaTeq, RotaTeq
Number analyzed (Participants) | 206 | 206 | 190 | 287 | 279
participants | 161 | 152 | 150 | 114 | 216

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited adverse events were collected for 8 days after each vaccination. Serious adverse events were collected from the first vaccination through the last follow-up visit at 6 months after the last vaccination.
Description: For events solicited on the memory aid in the 8 days after each vaccination, a participant was considered to have one event if it was reported as experienced at any time in the 8-day period. Each 8-day period was considered a separate event.
Arm/Group | Group 1: RotaTeq, RotaTeq, RotaTeq | Group 2: RotaTeq, Rotarix, Rotarix | Group 3: RotaTeq, RotaTeq, Rotarix | Group 4: Rotarix, Rotarix | Group 5: Rotarix, RotaTeq, RotaTeq
Serious Adverse Events (participants affected / at risk) | 11/242 | 7/248 | 13/238 | 11/329 | 21/327
Other Adverse Events (participants affected / at risk) | 75/242 | 95/248 | 98/238 | 85/329 | 135/327
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: RotaTeq, RotaTeq, RotaTeq (N=242) | Group 2: RotaTeq, Rotarix, Rotarix (N=248) | Group 3: RotaTeq, RotaTeq, Rotarix (N=238) | Group 4: Rotarix, Rotarix (N=329) | Group 5: Rotarix, RotaTeq, RotaTeq (N=327)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniosynostosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (5) | 0 (0) | 2 (2)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema herpeticum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulval cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gross motor delay (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: RotaTeq, RotaTeq, RotaTeq (N=242) | Group 2: RotaTeq, Rotarix, Rotarix (N=248) | Group 3: RotaTeq, RotaTeq, Rotarix (N=238) | Group 4: Rotarix, Rotarix (N=329) | Group 5: Rotarix, RotaTeq, RotaTeq (N=327)
Bronchiolitis (Infections and infestations) | 6 (6) | 11 (11) | 12 (14) | 3 (3) | 13 (15)
Irritability (General disorders) | 35 (44) | 38 (54) | 40 (51) | 53 (70) | 61 (90)
Otitis media (Infections and infestations) | 15 (17) | 14 (15) | 9 (11) | 4 (4) | 27 (29)
Pyrexia (General disorders) | 5 (5) | 9 (11) | 15 (15) | 6 (8) | 12 (13)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 13 (14) | 18 (18) | 7 (7) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 27 (29) | 38 (44) | 31 (34) | 24 (24) | 50 (61)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less